CLINICAL TRIAL: NCT02759536
Title: In-hospital Neutron Irradiator (IHNI)-Based Boron Neutron Capture Therapy (BNCT) in the Treatment of Malignant Melanoma: A Feasibility Study
Brief Title: In-hospital Neutron Irradiator (IHNI)-Based Boron Neutron Capture Therapy (BNCT) in the Treatment of Malignant Melanoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Collaborators: Beijing Capture Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XY3-IHNI1307A01
Record Dates: First submitted 2016-04-18; First posted 2016-05-03 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-04

CONDITIONS: Melanoma; Boron Neutron Capture Therapy
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Boronophenylalanine and IHNI-based BNCT (Experimental)
  Interventions: Radiation: Boronophenylalanine and IHNI-based BNCT

INTERVENTIONS:
Radiation: Boronophenylalanine and IHNI-based BNCT — Patients will be infused Boronophenylalanine (BPA)-fructose solution intravenously at a dose of 350mg/kg over 90 minutes. After BPA infusion, patients will receive neutron irradiation in IHNI for a certain period of time based on his boron bio-distribution curve and BPA concentration in the blood.

SUMMARY:
Boron Neutron Capture Therapy (BNCT) has been used in the treatment of several types of malignant tumors, including malignant melanoma, high-grade gliomas, and advanced head and neck cancers. Theoretically, it represents a more precise radiotherapy in that it could spare normal cells while destroy malignant ones. However, its value is largely restricted by the fact that it could only be performed in the nuclear research reactors, the only neutron source at the time. In 2010, the world's first in-hospital neutron irradiator (IHNI) had been constructed in Beijing, China, and this study aims to evaluate whether IHNI has the potential to serve as an effective in-hospital neutron source for BNCT.

DETAILED DESCRIPTION:
This is a single BNCT-facility, non-randomized, non-comparative, open-label, phase I to II clinical trial to determine the value of IHNI in the performance of BNCT. Before patients are recruited in this study, they must have been confirmed as malignant melanoma by biopsy and pathological analysis. Then they will receive a boron bio-distribution test, only patients whose boron concentration in tumor tissue is >1.5 times that in the blood will be enrolled. Before patients being irradiated in IHNI, they will be infused Boronophenylalanine (BPA)-fructose solution intravenously at a dose of 350mg/kg over 90 minutes, and then blood will be withdrawn from the patient at different time points to measure boron concentration. The start point and duration of irradiation will be determined based on the boron concentration in blood and the boron bio-distribution curve.

IHNI locates in Fangshan District, Beijing, China. The recruitment of patients, and their evaluation and medical care before and after BNCT will be done in the Third Xiangya Hospital, Changsha, China.

All patients will be evaluated for response by biopsy and pathological analysis, Positron Emission Computed Tomography (PET-CT), Computed Tomography (CT) or magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

1. Sign an informed consent form.
2. Age above 18, gender unlimited.
3. Expectation of life above 3 months.
4. Characteristic of disease: ① Pathological analysis confirms the diagnosis of melanoma. ② PET-CT and serum lactate dehydrogenase (LDH) can be used for auxiliary diagnosis. ③Diameter of at least one solid tumor ≥ 1cm.
5. KPS score: ≥70%.
6. Eastern Cooperative Oncology Group (ECOG) score: 0-2 grade.
7. (Within a week) Complete blood count: hemoglobin≥90g/L, leukocyte ≥ 4.0×109/L, neutrophilic granulocyte ≥ 2.0×109/L, platelet ≥ 100.0×109/L; Renal function: creatinine ≤ 180 umol/L.
8. Never accepted radiation or chemotherapy, or the interval of radiation or chemotherapy administered above 3 month.
9. Never accepted target drugs or biotherapeutics.
10. Urine pregnancy test negative (selectivity).

Exclusion Criteria:

1. Intolerable to BNCT treatment.
2. Sever coagulation disorders.
3. Poor compliance.
4. Sever complications or infection without control.
5. Pregnant woman or woman in lactation period.
6. Patients with metallic instruments (such as pacemaker, artificial limb).
7. Boron concentration in tumor tissue was <1.5 times that in blood.
8. Age<18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants showing CR/PR to IHNI-based BNCT | baseline and 2 years
  CT scan will be performed on each patient before and 2 years after irradiation, up to a maximum of 2 lesions of the longest diameter (unit: millimeter, mm) will be selected as target lesion(s). The diameter of the targeted lesion(s) will be measured on CT images. The change in the diameter of the targeted lesion(s) will be used to evaluate the patient's treatment response to IHNI-based BNCT according to Response Evaluation Criteria in Solid Tumors (RECIST). RECIST consists of four types of response: complete response (CR), partial response (PR), Stable Disease (SD), and Progressive Disease (PD). The percentage of participants who show CR/PR will be used to evaluate the efficiency of IHNI-based BNCT.

SECONDARY OUTCOMES:
Percentage of participants with treatment-related adverse events | 1 week, 1 month, 3 months, 6 months, 1 year and 2 years
  Physical examination, biochemical profile, routine blood test, and urine analysis will be performed on each patient at 1 week, 1 month, 3 months, 6 months, 1 year and 2 years after irradiation. All these results will be used to assess the grade of treatment-related adverse events according to Acute Radiation Morbidity Scoring Criteria and Late Radiation Morbidity Scoring Scheme from the Radiation Therapy Oncology Group (RTOG) and the European Organization for Research and Treatment of Cancer (EORTC). The percentage of adverse event at each grade will be used for the evaluation of the safety of IHNI-based BNCT.

OTHER OUTCOMES:
Percentage of participants of improved life quality. | baseline and 1 year
  This is to understand whether patients' life quality will be improved by BNCT, based on the Karnofsky performance status (KPS) score (unit: percentage, %) before and 1 year after irradiation. Questionnaires will be given to each patient at these two time points. The increase in KPS score after irradiation will be regarded as a reflection of improved life quality, and the percentage of participants who show improved life quality will be used to evaluate of benefits of IHNI-based BNCT.

CONTACTS AND LOCATIONS:
Overall Officials: Shaihong Zhu, M.D., Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ke G, Sun Z, Shen F, Liu T, Li Y, Zhou Y. The study of physics and thermal characteristics for in-hospital neutron irradiator (IHNI). Appl Radiat Isot. 2009 Jul;67(7-8 Suppl):S234-7. doi: 10.1016/j.apradiso.2009.03.117. Epub 2009 Apr 9. PMID 19427794